CLINICAL TRIAL: NCT03556150
Title: Effectiveness of a Manual Therapy Protocol in Patients With Masticatory Muscle Disorders: A Randomized Controlled Trial
Brief Title: Effectiveness of a Manual Therapy Protocol in Patients With Masticatory Muscle Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Beatriz Martín Bravo, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/HU/2018/05
Record Dates: First submitted 2018-06-02; First posted 2018-06-14 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Therapy protocol (Experimental): Massages, mobilisation and stretching techniques in the most painful joint
  Interventions: Other: Manual Therapy protocol
- Effleurage (Active Comparator): Superficial massage in the most painful joint.
  Interventions: Other: Effleurage

INTERVENTIONS:
Other: Manual Therapy protocol — This protocol consists of:
  * Six minutes of joint's mobilisation (two minutes of each technique).
  * Nine minutes of ischemic pressure . Three minutes per muscle in this order: temporal muscle, masseter muscle and lateral pterygoid. Choosing the two most painful trigger points.
  * Three minutes of trigemino's nerve stretching.
  Arms: Manual Therapy protocol
Other: Effleurage — The protocol consists of:
  * Five minutes in temporal muscle.
  * Ten minutes superficial massage in the neck and cheek of the most painful joint.
  * Five minutes of effleurage in the cheek, with the index finger inside the mouth and the thumb outside.
  Arms: Effleurage

SUMMARY:
Comparing the efficiency between manual therapy protocol and effleurage in patients with temporomandibular disorders.

DETAILED DESCRIPTION:
The investigators want to get better insights into the outcome of a manual therapy protocol compare with effleurage. The treatment is meant for people who has masticatory muscle disorders. Besides, if the trial can reduce the pain's intensity and the trial can improve range of motion in the dysfunction of temporomandibular joint. The results will be register on the short and long term.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are between 18 and 60 years old.
* Patients who have myofascial pain or myofascial pain and restricted oral opening taking into account Diagnostic Criteria for Temporomandibular Disorders (DC/TMD).
* Patients who have pain in their masticatory muscles while they are doing functional activities with their temporomandibular joint for, at least, the last six months.

Exclusion Criteria:

* Patients who cannot receive manual therapy.
* Patients who took or have been taking pills in the last two months before they start in the trial like: antidepressants, antiepileptics, muscle relaxants or medications for metabolic diseases; because they affect the musculoskeletal system.
* Surgery intervention in the temporomandibular joint.
* Patients who have received physiotherapy sessions in the last six months.
* Red flags: malignant or inflammatory tumors, infectious diseases that contraindicate manual therapy, cervical surgery, previous history of whiplash, fibromyalgia, trigeminal neuralgia, osteoarthritis or rheumatoid arthritis.
* Patients who lost their teeth (excluding the third molar) or people using a total or partial dentures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2018-09-03 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Measurements will be taken before the treatment starts, one hour after the last session, fifteen days after the last session and one month after the last session.
  It's an instrument to measure subjective pain intensity. It consists of a horizontal line of ten centimetres in length. On the left side appears the description of "no pain" and on the right side "the worst unimaginable pain". The patient is asked to draw a line at the point where he would place the intensity of his pain. Subsequently, it will be measured with a millimeter ruler from the left end to the point indicated by the patient. It will be the way to express in millimeters the intensity of pain. A minimum change of between 1.5 and 2.4 is required to be clinically significant, taking as reference the significant minimum change of subjects with nonspecific neck pain.
Oral opening | Measurements will be taken before the treatment starts, one hour after the last session, fifteen days after the last session and one month after the last session.
  It will use a rule of fifteen centimetres (starting from 0), to measure the maximum painless opening and the maximum total opening. The opening will be the measurement that is between the lower part of the incisors of the upper jaw and the upper part of the incisors of the lower jaw, not counting the vertical overbite. The patient will be asked to open their mouth as much as possible without pain and also as much as possible until their pain tolerance. It will be analyzed taking three measurements with a rest's interval of 30 seconds. The three measurements will be added up and the average will be taken to obtain the final result. The minimum detectable change to be clinically significant is 5 to 9 mm.
Pressure algometry measurement | Measurements will be taken before the treatment starts, one hour after the last session, fifteen days after the last session and one month after the last session.
  It measures the pain of the main masticatory muscles (temporal muscle, masseter muscle and lateral pterygoid muscle). The pain's pressure is analyzed three times at each point. The three measurements will be added up and the average will be taken to obtain the final result.
  The patient is in supine, the investigators apply the tip of the algometer perpendicular to the muscle maintaining a pressure, which will progressively increase up to 1kg / cm2. Participants will be instructed to make a nonverbal signal at the time they start to experience pain, in order to obtain an accurate record. The minimum detectable change to be clinically significant is 1.13kg / cm2, taking as reference the nonspecific neck pain.

SECONDARY OUTCOMES:
Self-perceived effect | Measurements will be taken one hour after the last session and one month after the last session.
  The effect and the level of patients' satisfaction will be measured, through a scale of 11 points. Patients will draw a circle depending on the change they have experienced from -5 (much worse), passing through 0 (unchanged) to the +5 (full recovery).

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz M. Bravo, Physiotherapy, Principal Investigator — Investigator; Inmaculada T. Tejada, Physiotherapy, Principal Investigator — Investigator
Locations (1):
- University of Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No